CLINICAL TRIAL: NCT03756363
Title: Postoperative Pain After Removal of Gutta-percha From Root Canals in Endodontic Retreatment Using a Solvent
Brief Title: The Effect of Solvent Usage on Post-treatment Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Ozgur Genc Sen, Assistant professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B.30.2.YYU.0.01.00.00/125
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Root Canal Infection; Pain
Keywords: Postoperative pain; Debris extrusion; Filling removal; solvent
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Solvents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-solvent (Experimental): Non-solvent use of a rotary retreatment system
  Interventions: Procedure: Non-solvent
- Solvent (Experimental): Solvent use in combination with a rotary retreatment system
  Interventions: Procedure: Solvent

INTERVENTIONS:
Procedure: Non-solvent — Root canal filling removal using ProTaper retreatment instruments. Single session retreatment procedures.
  Arms: Non-solvent
Procedure: Solvent — Root canal filling removal using ProTaper retreatment instruments in combination with a gutta percha solvent. Single session retreatment procedures.
  Arms: Solvent

SUMMARY:
No clinical evidence has been yet published regarding the comparison of postoperative pain after removal of the root canal fillings with or without solvent. The aim of this study was to evaluate the effect of combined usage of ProTaper retreatment instruments and a gutta-percha solvent, on the postoperative pain intensity after retreatment.

DETAILED DESCRIPTION:
Scientific literature contains a few studies regarding the amount of apically extruded debris caused by solvent or solvent free use of rotary instruments. It was reported that the use of ProTaper retreatment instruments in combination with gutta-percha solvent reduced the amount of apically extruded debris compared to their solvent free use. Nevertheless,no clinical evidence has been yet published regarding the comparison of postoperative pain after removal of the root canal fillings with or without solvent. The aim of this study was to evaluate the effect of combined usage of ProTaper retreatment instruments and gutta-percha solvent, on the postoperative pain intensity after retreatment. The adult patients (18-59 ages) who referred to Department of Endodontics with a diagnose of failed root canal treatment were examined radiographically and clinically. Endodontically treated, clinically asymptomatic, single-rooted teeth with one canal exhibiting chronic periapical infection were included. A hundred cases who matched the determined criteria were selected and randomly allocated to two groups:

Non-solvent Group (n=50):

ProTaper retreatment instruments were used in combination with with X-Smart electric motor for the removal of root canal fillings.

Solvent Group (n=50):

ProTaper retreatment instruments were used with the abovementioned technique but in combination with a gutta-percha solvent

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patient who has a failed root canal treatment.
* Asymptomatic single rooted teeth that had an initial root canal filling diagnosed with chronic apical periodontitis.
* Patients agreed to parcitipate in the study

Exclusion Criteria:

* Overfilled teeth,
* teeth with intraradicular posts,
* existence of a sinus tract,
* consumption of antibiotics or analgesics within one month,
* pregnancy,
* history of trauma,
* traumatic occlusion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-01-05 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after removal of gutta-percha with or without solvent | 24 hours postoperatively
  Pain intensity was evaluated at 24 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine'.All patients were requested to mark a number corresponding to their average pain.

SECONDARY OUTCOMES:
Postoperative pain after removal of gutta-percha with or without solvent | 24 to 48 hours postoperatively
  Pain intensity was evaluated at 48 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine' . All patients were requested to mark a number corresponding to their average pain.
Postoperative pain after removal of gutta-percha with or without solvent | 48 to 72 hours postoperatively
  Pain intensity was evaluated at 72 hours after retreatment procedures. An 11-item numerical rating scale (NRS) was used to assess the pain. This NRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0 -10 integers) that best reflects the intensity of their pain. Number 0 represents 'no pain' whereas number 10 represents 'pain as bad as someone can imagine'. All patients were requested to mark a number corresponding to their average pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur G Genc Sen, Principal Investigator — Yuzuncu Yil University, Faculty of Dentistry; Ali G Erdemir, Study Director — Yuzuncu Yil University, Faculty of Dentistry
Locations (1):
- Ozgur Genc Sen, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Genc Sen O, Erdemir A, Canakci BC. Effect of solvent use on postoperative pain in root canal retreatment: a randomized, controlled clinical trial. Clin Oral Investig. 2020 Jan;24(1):257-263. doi: 10.1007/s00784-019-02948-3. Epub 2019 May 15. PMID 31093742